CLINICAL TRIAL: NCT04444804
Title: Real-world Comparative Effectiveness of Rivaroxaban Versus Low-molecular-weight Heparin (LMWH) and Phenprocoumon for the Treatment and Secondary Prevention of Venous Thromboembolism (RECENT)
Brief Title: Study to Compare the Effectiveness of Rivaroxaban (Xarelto) Versus Low-molecular-weight Heparin (LMWH) and Phenprocoumon for the Treatment and Secondary Prevention of Venous Thromboembolism in Routine Clinical Practice in Germany
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21456
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Heparin, Low-Molecular-Weight; Phenprocoumon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rivaroxaban: The source population of this study will include all insured members of more than 60 German statutory health insurances (SHIs) contributing data to the InGef database.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY 59-7939)
- Low-molecular-weight heparin (LMWH) and Phenprocoumon: The source population of this study will include all insured members of more than 60 German statutory health insurances (SHIs) contributing data to the InGef database.
  Interventions: Drug: LMWH and Phenprocoumon

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY 59-7939) — Dosage at the discretion of the treating physician
  Groups: Rivaroxaban
Drug: LMWH and Phenprocoumon — Dosage at the discretion of the treating physician
  Groups: Low-molecular-weight heparin (LMWH) and Phenprocoumon

SUMMARY:
Researcher in this study want to compare the effectiveness of Rivaroxaban (Xarelto) versus low-molecular-weight heparin (LMWH) and phenprocoumon for the treatment and secondary prevention of venous thromboembolism by evaluating routine clinical practice data from research database in Germany. VTE is defined by a blood clot in the leg or lower extremity (deep vein thrombosis) or a blood clot in the lung (pulmonary embolism). Treatment of VTE traditionally consists of acute anticoagulation treatment with heparin (mainly LMWH), followed by maintenance oral anticoagulation with vitamin-K antagonists (in Germany mainly phenprocoumon). Rivaroxaban, a direct-acting oral anticoagulants (DOAC), is an alternative VTE treatment and has been approved for both the acute and maintenance phase of VTE treatment. The study will enroll adult male or female patients who are newly diagnosed with VTE and are already on the treatment with Rivaroxaban or LMWH and phenprocoumon. Researchers are especially interested whether patients experience under treatment any VTE events or fatal bleedings.

ELIGIBILITY:
Inclusion Criteria:

* At least one new diagnosis of VTE during the inclusion period:
* Ambulatory diagnosis, coded as verified,
* Primary hospital discharge diagnosis.
* Secondary hospital discharge diagnosis The quarter of the first VTE diagnosis in the inclusion period will be defined as the index quarter. For hospital diagnoses, the date of admission will be used to define the index quarter.
* The 12 months prior to the index date will define the baseline period for all included patients. Patients treated with anticoagulation regimens other than defined above (e.g. other DOACs) will not be included in the study. All patients will have to fulfill the additional inclusion criteria:
* Continuous enrolment in the baseline period
* ≥ 18 years of age at index date

Exclusion Criteria:

* A verified ambulatory or primary/ secondary hospital discharge diagnosis of VTE in the baseline period;
* A verified ambulatory or primary/ secondary hospital discharge diagnosis of atrial fibrillation in the baseline period; Individuals with documented cardiac valve surgery in the baseline period;
* A verified ambulatory or primary/ secondary hospital discharge diagnosis indicating pregnancy in the baseline period;
* A prescription of any anticoagulation treatment (heparins; vitamin-K antagonists; rivaroxaban; other DOACs) in the baseline period;
* A verified ambulatory or primary/ secondary hospital discharge diagnosis of end-stage kidney disease or a claim for dialysis in the baseline period;
* A prescription of contraindicated drug for rivaroxaban due to drug interactions (i.e. azole antifungals and HIV protease inhibitors) in the 60 days before or on the index date.
* Patients assigned to rivaroxaban exposure groups who were initially treated with a dose strength other than 15 mg or 20 mg per tablet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The source population of this study will include all insured members of more than 60 German statutory health insurances (SHIs) contributing data to the InGef database.
Sampling Method: Non-Probability Sample
Enrollment: 22153 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Risk of recurrent venous thromboembolic (VTE) events in VTE patients treated with rivaroxaban compared to patients treated with LMWH and Phenprocoumon | Retrospective data from January 2013 to December 2018
  A recurrent VTE event will be defined as a hospitalization with a primary hospital discharge diagnoses for VTE for which the admission date was >14 days after the index date.
  Non-interventional retrospective cohort study based on German claims data from the InGef (Institute for Applied Healthcare Research Berlin) research database between January 2013 and December 2018.

SECONDARY OUTCOMES:
Risk of fatal bleeding in VTE patients treated with rivaroxaban compared to patients treated with LMWH and Phenprocoumon | Retrospective data from January 2013 to December 2018
  Cases of fatal bleeding will be defined as hospitalization with a primary hospital discharge diagnoses for bleeding with documented death as reason for hospital discharge or within 30 days after hospital discharge.
  Non-interventional retrospective cohort study based on German claims data from the InGef (Institute for Applied Healthcare Research Berlin) research database between January 2013 and December 2018.

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple facilities, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.